CLINICAL TRIAL: NCT03037528
Title: Examination of Psychological Tools and Tracking in an Online Intervention for Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Laura Saslow, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00115537; 5K01DK107456-05 (NIH)
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Diet

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Positive Affect, Mindfulness, Tracking (Experimental): Participants will receive information about positive affect and mindfulness, in addition to being asked to actively track what they eat and receiving the core program
  Interventions: Behavioral: diet and lifestyle program; Behavioral: positive affect informational materials; Behavioral: mindfulness informational materials; Behavioral: dietary tracking
- Mindfulness, Tracking (Experimental): Participants will receive information about mindfulness, be asked to actively track what they eat, and receive the core program.
  Interventions: Behavioral: diet and lifestyle program; Behavioral: mindfulness informational materials; Behavioral: dietary tracking
- Positive Affect, Tracking (Experimental): Participants will receive information about positive affect, be asked to actively track what they eat, and receive the core program.
  Interventions: Behavioral: diet and lifestyle program; Behavioral: positive affect informational materials; Behavioral: dietary tracking
- Tracking (Experimental): Participants will be asked to actively track what they eat in addition to receiving the core program.
  Interventions: Behavioral: diet and lifestyle program; Behavioral: dietary tracking
- Positive Affect, Mindfulness (Experimental): Participants will receive information about positive affect and mindfulness in addition to the core program.
  Interventions: Behavioral: diet and lifestyle program; Behavioral: positive affect informational materials; Behavioral: mindfulness informational materials
- Positive Affect (Experimental): Participants will receive information about positive affect in addition to the core program.
  Interventions: Behavioral: diet and lifestyle program; Behavioral: positive affect informational materials
- Mindfulness (Experimental): Participants will receive information about mindfulness in addition to the core program.
  Interventions: Behavioral: diet and lifestyle program; Behavioral: mindfulness informational materials
- No Extras (Experimental): Participants will receive the core program.
  Interventions: Behavioral: diet and lifestyle program

INTERVENTIONS:
Behavioral: diet and lifestyle program — Participants will be taught how to follow a very low carbohydrate, ketogenic diet, become more physically active, and get adequate sleep.
Behavioral: positive affect informational materials — Participants will be taught about positive affect skills, such as gratitude, positive reappraisal, and personal strengths.
  Arms: Positive Affect; Positive Affect, Mindfulness; Positive Affect, Mindfulness, Tracking; Positive Affect, Tracking
Behavioral: mindfulness informational materials — Participants will be taught about mindfulness and mindful eating techniques.
  Arms: Mindfulness; Mindfulness, Tracking; Positive Affect, Mindfulness; Positive Affect, Mindfulness, Tracking
Behavioral: dietary tracking — Participants will be asked to track their diet consistently.
  Arms: Mindfulness, Tracking; Positive Affect, Mindfulness, Tracking; Positive Affect, Tracking; Tracking

SUMMARY:
The goal of the research is to optimize an online and mobile multicomponent 12-month diet and lifestyle intervention for improving the blood glucose control of individuals with type 2 diabetes.

DETAILED DESCRIPTION:
The core of the program, administered to all participants, includes recommendations to follow a very low carbohydrate, ketogenic diet. The researchers will test whether adding the following experimental components will enhance the intervention's ability to improve health outcomes: (1) active vs. periodic self-monitoring of dietary intake using an "app"; (2) training vs. no training in positive affect; and (3) training vs. no training in mindfulness and mindful eating.

ELIGIBILITY:
Inclusion Criteria:

* Weight: Body Mass Index of 25-45 kg/m2 or greater.
* Current HbA1c of 6.5% or higher
* Regular access to the internet

Exclusion Criteria:

* Taking glucose lowering medications other than metformin
* Being pregnant or breastfeeding
* Currently undergoing cancer treatments
* Active use of a weight loss program or medications
* Self-reported impaired renal or hepatic function
* Self-reported untreated thyroid condition
* Vegetarian or vegan
* Weight loss surgery within the past year
* Medical concerns that prevent participants from following the assigned protocol

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saslow LR, Missel AL, O'Brien A, Kim S, Hecht FM, Moskowitz JT, Bayandorian H, Pietrucha M, Raymond K, Richards B, Liestenfeltz B, Mason AE, Daubenmier J, Aikens JE. Psychological Support Strategies for Adults With Type 2 Diabetes in a Very Low-Carbohydrate Web-Based Program: Randomized Controlled Trial. JMIR Diabetes. 2023 May 11;8:e44295. doi: 10.2196/44295. PMID 37166961

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited 112 participants.
Pre-assignment Details: In this 2x2x2 design, rather than considering this as an 8-arm trial, we consider this a trial assessing 3 factors at two levels, and we compare each of the 3 factors, rather than comparing the study arms.
Groups:
- Positive Affect, Mindfulness, and Daily Tracking: Participants were assigned to Positive affect, Mindfulness, and Daily Tracking
- Mindfulness and Daily Tracking: Participants were assigned to Mindfulness and Daily Tracking
- Positive Affect and Daily Tracking: Participants were assigned to Positive Affect and Daily Tracking
- Daily Tracking: Participants were assigned to Daily Tracking
- Positive Affect, Mindfulness, Monthly Tracking: Participants were assigned to Positive Affect, Mindfulness, Monthly Tracking
- Mindfulness and Monthly Tracking: Participants were assigned to Mindfulness and Monthly Tracking
- Positive Affect and Monthly Tracking: Participants were assigned to Positive Affect and Monthly Tracking
- Monthly Tracking: Participants were assigned to Monthly Tracking
Period: Overall Study
Arm/Group | Positive Affect, Mindfulness, and Daily Tracking | Mindfulness and Daily Tracking | Positive Affect and Daily Tracking | Daily Tracking | Positive Affect, Mindfulness, Monthly Tracking | Mindfulness and Monthly Tracking | Positive Affect and Monthly Tracking | Monthly Tracking
Started | 15 | 15 | 13 | 14 | 13 | 14 | 15 | 13
Completed | 12 | 12 | 11 | 10 | 8 | 7 | 9 | 5
Not Completed | 3 | 3 | 2 | 4 | 5 | 7 | 6 | 8

BASELINE CHARACTERISTICS:
Groups:
- Positive Affect, Mindfulness, and Daily Tracking: Diet and Lifestyle Program: Participants will be taught how to follow a very low carbohydrate, ketogenic diet, become more physically active, and get adequate sleep.
  Positive Affect, Mindfulness, and Daily Tracking:
  positive affect informational materials (yes): Participants will be taught about positive affect skills, such as gratitude, positive reappraisal, and personal strengths.
  mindfulness informational materials (yes): Participants will be taught about mindfulness and mindful eating techniques.
  dietary tracking (daily): Participants will be asked to track their diet daily.
- Mindfulness and Daily Tracking: Diet and Lifestyle Program: Participants will be taught how to follow a very low carbohydrate, ketogenic diet, become more physically active, and get adequate sleep.
  mindfulness informational materials (yes): Participants will be taught about mindfulness and mindful eating techniques.
  dietary tracking (daily): Participants will be asked to track their diet daily.
- Positive Affect and Daily Tracking: Diet and Lifestyle Program: Participants will be taught how to follow a very low carbohydrate, ketogenic diet, become more physically active, and get adequate sleep.
  positive affect informational materials (yes): Participants will be taught about positive affect skills, such as gratitude, positive reappraisal, and personal strengths.
  dietary tracking (daily): Participants will be asked to track their diet daily.
- Daily Tracking: Diet and Lifestyle Program: Participants will be taught how to follow a very low carbohydrate, ketogenic diet, become more physically active, and get adequate sleep.
  dietary tracking (daily): Participants will be asked to track their diet daily.
- Positive Affect, Mindfulness, Monthly Tracking: Diet and Lifestyle Program: Participants will be taught how to follow a very low carbohydrate, ketogenic diet, become more physically active, and get adequate sleep.
  positive affect informational materials (yes): Participants will be taught about positive affect skills, such as gratitude, positive reappraisal, and personal strengths.
  mindfulness informational materials (yes): Participants will be taught about mindfulness and mindful eating techniques.
  dietary tracking (monthly): Participants will be asked to track their diet monthly.
- Mindfulness and Monthly Tracking: Diet and Lifestyle Program: Participants will be taught how to follow a very low carbohydrate, ketogenic diet, become more physically active, and get adequate sleep.
  mindfulness informational materials (yes): Participants will be taught about mindfulness and mindful eating techniques.
  dietary tracking (monthly): Participants will be asked to track their diet monthly.
- Positive Affect and Monthly Tracking: Diet and Lifestyle Program: Participants will be taught how to follow a very low carbohydrate, ketogenic diet, become more physically active, and get adequate sleep.
  positive affect informational materials (yes): Participants will be taught about positive affect skills, such as gratitude, positive reappraisal, and personal strengths.
  dietary tracking (monthly): Participants will be asked to track their diet monthly.
- Monthly Tracking: Diet and Lifestyle Program: Participants will be taught how to follow a very low carbohydrate, ketogenic diet, become more physically active, and get adequate sleep.
  dietary tracking (monthly): Participants will be asked to track their diet monthly.
- Total: Total of all reporting groups
Arm/Group | Positive Affect, Mindfulness, and Daily Tracking | Mindfulness and Daily Tracking | Positive Affect and Daily Tracking | Daily Tracking | Positive Affect, Mindfulness, Monthly Tracking | Mindfulness and Monthly Tracking | Positive Affect and Monthly Tracking | Monthly Tracking | Total
Number analyzed (Participants) | 15 | 15 | 13 | 14 | 13 | 14 | 15 | 13 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (10.7) | 50.2 (8.9) | 53.4 (11.3) | 54.9 (11.0) | 55.9 (6.6) | 55.9 (9.6) | 58.0 (7.0) | 53.0 (11.1) | 54.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 10 | 10 | 10 | 10 | 11 | 10 | 83
  Male | 4 | 4 | 3 | 4 | 3 | 4 | 4 | 3 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 15 | 13 | 14 | 13 | 14 | 14 | 13 | 111
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 10 | 9 | 11 | 9 | 13 | 9 | 9 | 81
  African American | 4 | 4 | 3 | 3 | 3 | 1 | 5 | 4 | 27
  Other | 0 | 2 | 1 | 0 | 2 | 0 | 1 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Glycemic Control
Description: Measured with HbA1c
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: change in units of percents
Groups:
- Positive Affect, Mindfulness, and Daily Tracking: Diet and Lifestyle Program: Participants will be taught how to follow a very low carbohydrate, ketogenic diet, become more physically active, and get adequate sleep.
  positive affect informational materials (yes): Participants will be taught about positive affect skills, such as gratitude, positive reappraisal, and personal strengths.
  mindfulness informational materials (yes): Participants will be taught about mindfulness and mindful eating techniques.
  dietary tracking (daily): Participants will be asked to track their diet daily.
Arm/Group | Positive Affect, Mindfulness, and Daily Tracking | Mindfulness and Daily Tracking | Positive Affect and Daily Tracking | Daily Tracking | Positive Affect, Mindfulness, Monthly Tracking | Mindfulness and Monthly Tracking | Positive Affect and Monthly Tracking | Monthly Tracking
Number analyzed (Participants) | 12 | 12 | 11 | 10 | 8 | 7 | 9 | 5
change in units of percents | -.46 (1.20) | -.93 (1.14) | -.46 (1.99) | -.23 (1.27) | -1.23 (2.93) | -1.34 (0.61) | -.58 (0.48) | -.64 (0.78)
Statistical Analysis 1: Comparison: Positive Affect, Mindfulness, and Daily Tracking; Test type: Superiority; p = .214, t-test, 2 sided
Statistical Analysis 2: Comparison: Mindfulness and Daily Tracking; Test type: Superiority; p = .017, t-test, 2 sided
Statistical Analysis 3: Comparison: Positive Affect and Daily Tracking; Test type: Superiority; p = .457, t-test, 2 sided
Statistical Analysis 4: Comparison: Daily Tracking; Test type: Superiority; p = .580, t-test, 2 sided
Statistical Analysis 5: Comparison: Positive Affect, Mindfulness, Monthly Tracking; Test type: Superiority; p = .275, t-test, 2 sided
Statistical Analysis 6: Comparison: Mindfulness and Monthly Tracking; Test type: Superiority; p = .001, t-test, 2 sided
Statistical Analysis 7: Comparison: Positive Affect and Monthly Tracking; Test type: Superiority; p = .007, t-test, 2 sided
Statistical Analysis 8: Comparison: Monthly Tracking; Test type: Superiority; p = .142, t-test, 2 sided

2. Secondary Outcome: Weight Loss
Description: Measured with percent change in body weight
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: change in percent
Arm/Group | Positive Affect, Mindfulness, and Daily Tracking | Mindfulness and Daily Tracking | Positive Affect and Daily Tracking | Daily Tracking | Positive Affect, Mindfulness, Monthly Tracking | Mindfulness and Monthly Tracking | Positive Affect and Monthly Tracking | Monthly Tracking
Number analyzed (Participants) | 12 | 12 | 12 | 11 | 8 | 8 | 9 | 5
change in percent | -5.69 (8.03) | -9.60 (7.16) | -10.00 (14.80) | -5.25 (5.94) | -9.14 (8.33) | -9.85 (11.28) | -10.05 (10.27) | -3.84 (4.92)
Statistical Analysis 1: Comparison: Positive Affect, Mindfulness, and Daily Tracking; Test type: Superiority; p = .027, t-test, 2 sided
Statistical Analysis 2: Comparison: Mindfulness and Daily Tracking; Test type: Superiority; p = .000, t-test, 2 sided
Statistical Analysis 3: Comparison: Positive Affect and Daily Tracking; Test type: Superiority; p = .054, t-test, 2 sided
Statistical Analysis 4: Comparison: Daily Tracking; Test type: Superiority; p = .014, t-test, 2 sided
Statistical Analysis 5: Comparison: Positive Affect, Mindfulness, Monthly Tracking; Test type: Superiority; p = .019, t-test, 2 sided
Statistical Analysis 6: Comparison: Mindfulness and Monthly Tracking; Test type: Superiority; p = .026, t-test, 2 sided
Statistical Analysis 7: Comparison: Positive Affect and Monthly Tracking; Test type: Superiority; p = .013, t-test, 2 sided
Statistical Analysis 8: Comparison: Monthly Tracking; Test type: Superiority; p = .163, t-test, 2 sided

3. Secondary Outcome: Depressive Symptoms
Description: Measured with Patient Health Questionnaire-8. Eight items, each of which is scored 0 to 3, for a 0 to 24 severity score, with higher being a worse outcome.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Positive Affect, Mindfulness, and Daily Tracking | Mindfulness and Daily Tracking | Positive Affect and Daily Tracking | Daily Tracking | Positive Affect, Mindfulness, Monthly Tracking | Mindfulness and Monthly Tracking | Positive Affect and Monthly Tracking | Monthly Tracking
Number analyzed (Participants) | 12 | 10 | 10 | 11 | 8 | 7 | 8 | 5
units on a scale | -2.50 (3.12) | -2.70 (2.26) | -4.00 (7.67) | 0.00 (1.90) | -3.38 (4.00) | -3.71 (4.39) | -5.86 (6.15) | -4.60 (3.78)
Statistical Analysis 1: Comparison: Positive Affect, Mindfulness, and Daily Tracking; Test type: Superiority; p = .018, t-test, 2 sided
Statistical Analysis 2: Comparison: Mindfulness and Daily Tracking; Test type: Superiority; p = .004, t-test, 2 sided
Statistical Analysis 3: Comparison: Positive Affect and Daily Tracking; Test type: Superiority; p = .134, t-test, 2 sided
Statistical Analysis 4: Comparison: Daily Tracking; Test type: Superiority; p = 1.000, t-test, 2 sided
Statistical Analysis 5: Comparison: Positive Affect, Mindfulness, Monthly Tracking; Test type: Superiority; p = .048, t-test, 2 sided
Statistical Analysis 6: Comparison: Mindfulness and Monthly Tracking; Test type: Superiority; p = .066, t-test, 2 sided
Statistical Analysis 7: Comparison: Positive Affect and Monthly Tracking; Test type: Superiority; p = .045, t-test, 2 sided
Statistical Analysis 8: Comparison: Monthly Tracking; Test type: Superiority; p = .053, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: The entire course of the trial (12 months).
Description: This was a low-risk trial.
Arm/Group | Positive Affect, Mindfulness, and Daily Tracking | Mindfulness and Daily Tracking | Positive Affect and Daily Tracking | Daily Tracking | Positive Affect, Mindfulness, Monthly Tracking | Mindfulness and Monthly Tracking | Positive Affect and Monthly Tracking | Monthly Tracking
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/13 | 0/14 | 0/13 | 0/14 | 0/15 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/13 | 0/14 | 0/13 | 0/14 | 0/15 | 0/13
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/13 | 0/14 | 0/13 | 0/14 | 0/15 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-01-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT03037528/Prot_SAP_ICF_000.pdf